CLINICAL TRIAL: NCT02227368
Title: A Phase II Multicentre, Randomised, Double-Blind, Controlled, Parallel-Group Study to Evaluate the Walking Time Effect of Long-Term Ticagrelor in Comparison to Long-Term Aspirin Administration in Ambulatory Patients With Peripheral Artery Disease Undergoing Endovascular Revascularization - The Ticagrelor in Peripheral Artery Disease Endovascular Revascularization Study TI-PAD I EVR
Brief Title: Walking Effect of Long Term Ticagrelor in Subjects With PAD Who Have Undergone EVR
Acronym: TI-PAD EVR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: CPC Clinical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5135L00003
Record Dates: First submitted 2014-08-19; First posted 2014-08-28 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Peripheral Artery Disease (PAD)
Keywords: Myocardial Infarction; Peripheral Arterial disease; Mycardial Ischemia; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Altherosclerosis; Arteriosclerosis; Arterial Occlusive Diseases; Peripheral Vascular Diseases; Ticagrelor; Ticlopidine; Platelet Aggregation inhibitors; Hematologic Agents; Therapeutic Uses; Pharmacologic Actions; Purinegic P2Y Receptor Antagonists; Purinegic P2 Receptor Antagonists; Purinergic Antagonists; Purinergic Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Actions; Physiological Effects of Drugs; Fibrinolytic Agents; Crardiovascular Agents
MeSH Terms: conditions — Peripheral Arterial Disease; Myocardial Infarction; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Peripheral Vascular Diseases | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): 26 Weeks of ticagrelor 90mg twice a day plus aspirin placebo once daily
  Interventions: Drug: Ticagrelor
- Aspirin (Active Comparator): 26 Weeks of aspirin 100mg once daily plus ticagrelor placebo twice a day
  Interventions: Drug: Comparator

INTERVENTIONS:
Drug: Ticagrelor — Antiplatelet therapy approved for ACS. Antagonist of P2Y12 and inhibitor of adenosine diphosphate (ADP)-induced platelet aggregation.
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Comparator — Aspirin monotherapy anti-platelet treatment for PAD patients following EVR procedures
  Other Names: Aspirin
  Arms: Aspirin

SUMMARY:
To compare the effect of ticagrelor versus aspirin on the change in peak walking time, evaluated on the graded treadmill test, from one to 26 weeks post-revascularization in patients with peripheral artery disease who have undergone endovascular revascularization for moderate to severe claudication or ischemic rest pain.

DETAILED DESCRIPTION:
A Phase II Multicentre, Randomised, Double-Blind, Controlled, Parallel-Group Study to Evaluate the Walking Time Effect of Long-Term Ticagrelor in Comparison to Long-Term Aspirin Administration in Ambulatory Patients with Peripheral Artery Disease Undergoing Endovascular Revascularization - The Ticagrelor in Peripheral Artery Disease Endovascular Revascularization Study TI-PAD I EVR.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent prior to any study specific procedures.
2. Ambulatory male or female outpatients aged 50 years of age or older at the time of the Screening Visit.
3. EVR, below the inguinal ligament that includes the distal SFA and/or popliteal and/or tibial arteries, that is planned to occur within 5 weeks after the Screening Visit, as determined and clearly documented by the Principal Investigator or physician Sub-Investigator (MD/DO). Patients undergoing a proximal revascularization may be enrolled as long as their procedure also includes treating the distal SFA, popliteal or tibial arteries. The EVR must be confirmed as technically successful (a completed procedure where haemostasis has been achieved) before the patient is randomised.
4. Normal inflow into the lower extremity as determined by the Principal Investigator or physician Sub-Investigator (MD/DO). Adequacy of inflow can be assessed by hemodynamic measures, angiography or other imaging modalities obtained during Screening or recorded in the medical records up to 30 days prior to the Screening Visit or as defined by imaging at the time of the procedure. A patient with inadequate inflow at the time of Screening can still be enrolled if the inflow is addressed and resolved by the planned revascularization procedure.
5. Diagnosis of PAD confirmed by history and any one of the following observed in the index (intervention) leg at the Screening Visit:

   1. Resting ABI ≤0.90, or
   2. In patients with an ABI > 1.40 (non-compressible vessels) a resting GTI <0.70 can be used for inclusions.
6. Patient has been advised of the beneficial effects of smoking cessation and exercise therapy but is not in the process of changing their smoking status or exercise at the time of the Screening Visit.

Exclusion Criteria

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Revascularisation planned only to treat proximal (inflow) disease in the iliac and/or common femoral arteries.
3. Previous randomisation in the present study.
4. Participation in another clinical study with an investigational product within the last 3 months or any new clinical trial during the course of this study.
5. Gangrene or ischemic ulcer of either lower extremity.
6. PAD of a non-atherosclerotic nature.
7. Clinical necessity to use dual antiplatelet therapy within 7 days prior to randomisation, or single anti-platelet therapy (ticlopidine, prasugrel, vorapaxar, ticagrelor or dipyridamole) other than clopidogrel or aspirin. Clopidogrel or aspirin can be taken up to and including the time that the loading dose is being given.
8. Clinical necessity to use the following restricted concomitant medications within 4 weeks prior to randomisation. Patients taking any of these medications at the Screening Visit may be considered for randomisation after a 4 week washout period from the medication.

   1. Pentoxifylline or cilostazol for relief of claudication symptoms
   2. Chronic oral or parenteral anticoagulant therapy (greater than 7 days)
   3. Strong inhibitors of CYP3A enzymes (Section 5.6.9.1)
   4. Strong inducers of CYP3A enzymes (Section 5.6.9.2)
   5. Simvastatin or lovastatin at daily doses over 40 mg
9. Any disease process (e.g. angina, cardiac abnormality, congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD), respiratory disease, obesity, stroke, severe neuropathy of the foot, symptomatic musculoskeletal disease of the lower extremity), other than PAD, that would interfere with exercise performance during the ETT or prevent the patient from reaching their claudication-limited PWT as the primary endpoint of the study.
10. Coronary, aortic surgery, angioplasty, lumbar sympathectomy or lower extremity surgery that impacts the ability to walk on a treadmill within the past 3 months prior to EVR. Revascularization of the non-index lower extremity within the past 4 weeks prior to EVR.
11. Any major lower limb amputation due to PAD anticipated within the next 3 months or prior major amputation due to PAD (minor toe amputations allowed if it does not interfere with ambulation).
12. Myocardial infarction or stroke in the previous 3 months.
13. Any concomitant disease process with a life expectancy of less than 1 year or which is sufficiently severe as to compromise the validity of test performance.
14. Dementia likely to jeopardise understanding of information pertinent to study conduct or compliance to study procedures.
15. Concern for the inability of the patient to comply with study procedures and/or followup (e.g., alcohol or drug abuse).
16. Resting systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥95 mmHg at the Screening Visit, in spite of antihypertensive treatments allowed by the protocol.
17. A known bleeding diathesis, haemostatic or coagulation disorder, or systemic bleeding, whether resolved or ongoing.
18. Known severe liver disease (e.g., ascites and or clinical signs of coagulopathy).
19. Renal failure requiring dialysis.
20. History of previous intracranial bleed at any time, gastrointestinal bleed within the past 6 months, or major surgery within 30 days (if the surgical wound is judged to be associated with an increased risk of bleeding).
21. History of thrombocytopenia or neutropenia.
22. Hypersensitivity to ticagrelor, aspirin or lactose.
23. Initiation of antidiabetic, antihypertensive, lipid-lowering and beta-blocking drugs within 1 month prior to the Screening Visit.
24. Pregnancy, lactation, fertility without protection against pregnancy (for women of childbearing potential; a urine or serum pregnancy test will be performed at the Screening Visit).

Ages: 50 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2016-05-23 (Actual); Study Completion 2016-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Hiatt, MD, Principal Investigator — Colorado Prevention Center Clinical Research
Locations (10):
- United States (10):
  - Research Site, Daytona Beach, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Ocala, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Munster, Indiana
  - Research Site, New York, New York
  - Research Site, Yonkers, New York
  - Research Site, Cleveland, Ohio
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas

REFERENCES:
- [Derived] Rogers RK, Hiatt WR, Patel MR, Shishehbor MH, White R, Khan ND, Bhalla NP, Jones WS, Low Wang CC. Ticagrelor in Peripheral Artery Disease Endovascular Revascularization (TI-PAD): Challenges in clinical trial execution. Vasc Med. 2018 Dec;23(6):513-522. doi: 10.1177/1358863X18760996. Epub 2018 Apr 9. PMID 29629845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 71 subjects were screened at 16 centers throughout the United States of America (USA).
  First subject enrolled: 20Oct2014. Last subject last visit: 23May2016. Date of early study termination: 21Oct2015
Pre-assignment Details: A total of 40 subjects were randomised. Thirty-one subjects were not randomised due to not meeting inclusion/exclusion criteria (20 subjects), withdrawing consent prior to randomisation (2 subjects), and other reasons (9 subjects) including not being able to return for randomisation within 48 hours of the qualifying revascularization.
Groups:
- Ticagrelor: Ticagrelor 90mg twice a day plus aspirin placebo once daily
- Aspirin: Aspirin 100mg once daily plus ticagrelor placebo twice a day
Period: Overall Study
Arm/Group | Ticagrelor | Aspirin
Started | 16 | 24
Sujects Who Received Treatment | 16 | 24
Sujects Who Completed Treatment | 10 | 17
Completed | 14 (Subjects who discontinued treatment were encouraged to remain in the study.) | 20 (Subjects who discontinued treatment were encouraged to remain in the study.)
Not Completed | 2 | 4
Not completed — No EVR/not PAD/PI decision/RLE bypass | 0 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomised subjects with the exception of one subject who did not undergo EVR.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Aspirin | Total
Number analyzed (Participants) | 16 | 24 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (9.15) | 67.0 (8.31) | 67.9 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 7 | 15 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 13 | 21 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 11 | 20 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log Transformed Peak Walking Time (PWT) at Week 26 or Early Termination (ET)
Time Frame: 26 Weeks
Population: ITT population is the analysis population. Six subjects without evaluable baseline were excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: log(Second)
Arm/Group | Ticagrelor | Aspirin
Number analyzed (Participants) | 14 | 20
log(Second) | 0.0 [-0.2 to 0.2] | 0.1 [-0.0 to 0.3]
Statistical Analysis 1: Comparison: Ticagrelor vs Aspirin; Test type: Superiority or Other; p = 0.3441, t-test, 2 sided; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.1] — Difference is Ticagrelor - Aspirin. LOCF was used for missing data imputation

2. Secondary Outcome: Change From Baseline in Log Transformed Claudication Onset Time (COT) at Week 26 or Early Termination (ET)
Time Frame: 26 Weeks
Population: ITT population is the analysis population. Twelve subjects without evaluable baseline were excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: log(Second)
Arm/Group | Ticagrelor | Aspirin
Number analyzed (Participants) | 12 | 16
log(Second) | 0.6 [0.1 to 1.1] | 0.5 [0.1 to 0.8]
Statistical Analysis 1: Comparison: Ticagrelor vs Aspirin; Test type: Superiority or Other; p = 0.6186, t-test, 2 sided; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.4 to 0.6] — Difference is Ticagrelor - Aspirin. LOCF was used for missing data imputation

ADVERSE EVENTS:
Time Frame: 26 weeks treatment period + 30 days followup
Description: Only SAEs and AEs of interest were collected for this study. Treatment Emergent SAEs and Treatment Emergent AEs of interest are reported here.
Arm/Group | Ticagrelor | Aspirin
Serious Adverse Events (participants affected / at risk) | 4/16 | 2/24
Other Adverse Events (participants affected / at risk) | 1/16 | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor (N=16) | Aspirin (N=24)
Coronary artery disease (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor (N=16) | Aspirin (N=24)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early for low enrolment. Less than 25% of anticipated number of subjects were enroled and there was an imbanlance between groups. Therefore, the results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require Confidential Information to be removed and the sponsor can extend the embargo for an additional 90 days.